# Participatory Research for Suicide Prevention in Autism

NCT06552871

Principal Investigator: Anne Kirby

Document date: 2024-07-08

## Study Protocol and Statistical Analysis Plan – Aim 3 (Clinical Trial)

## **Study Protocol**

Single arm, pre-test post-test pilot study of the Forming Love around Autistic people to Prevent Suicide (FLAPS) intervention.

#### Recruitment

We will recruit participants for FLAPS by first reaching out to organizations and inviting an organization representative to complete an interest form.

Once an organization agrees to participate, the organization representative will send out individual-level recruitment invitations to others in their organization with a link to consent information and a baseline study survey administered through Qualtrics. Via the survey, participants will be provided more information about the study and determine if they will participate in the program with their organization and consent to enroll in the study. The survey will collect participant-level descriptive information, baseline questionnaire data, contact information, and accessibility needs.

Upon completion of the study, participants will receive a gift card of up to \$70, prorated based on the study components they completed.

# **Program Implementation**

We will implement the group-based FLAPS program virtually over Zoom in sets of four 2-hour sessions. We sent log-on information and schedule reminders to each participant via email. After each session, we will provide all participants with additional program resources.

#### **Data Collection**

To measure the short-term outcomes of FLAPS (i.e., suicide prevention knowledge, capacity, and actions), we adapted the Steps Toward Prevention (STP) questionnaire (from Wexler et al., 2025; PMC11980237). The AASPIRE SPP team adapted the STP to align with the focus of FLAPS, creating the STP-Autism Community Suicide Prevention questionnaire. The STP-Autism Community Suicide Prevention questionnaire includes items on knowledge, capacity, and actions related to suicide prevention in general as well as specific to the autistic community.

In the post-program survey, participants will be asked to rate their satisfaction with the program. We will collect additional information about program relevance and application of program information in their organization. Optional post-program qualitative interviews will be conducted by a research team member who was not involved with implementation.

#### **Statistical Analysis Plan**

We will calculate descriptive statistics for participant demographics, descriptive information, and scaled feedback items.

We will also apply descriptive statistics to summarize data collected about engagement and participation in the program.

For the primary outcomes on the STP-Autism Community Suicide Prevention questionnaire, we will first examine the individual-level means and standard deviations on the average scores for each construct at all three timepoints using t-tests and Cohen's D effect sizes. Then we will conduct multi-level generalized linear models using baseline-observation-carried-forward technique and accounting for nesting within organizations.